CLINICAL TRIAL: NCT05449860
Title: Radiofrequency Ablation for Recurrent Hepatocellular Carcinoma After Locoregional Treatment Using Combined Bipolar and Monopolar Energy Deliver With Twin Cooled-Wet Electrodes: A Prospective Observational Study
Brief Title: Radiofrequency Ablation for Recurrent Hepatocellular Carcinoma With Twin Cooled-wet Electrodes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: RF medical (Unknown)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1907-157-1050
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma; Local Recurrence of Malignant Tumor of Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with recurrent hepatocellular carcinoma after locoregional treatment (Experimental): Patients with chronic liver disease have recurrent hepatocellular carcinoma which is diagnosed on contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI).
  Interventions: Procedure: Radiofrequency ablation using combined bipolar and monopolar energy deliver with Twin Cooled-Wet electrodes

INTERVENTIONS:
Procedure: Radiofrequency ablation using combined bipolar and monopolar energy deliver with Twin Cooled-Wet electrodes — Radiofrequency ablation will be performed by using twin cooled-wet electrodes. Two electrodes will be places on the tumor under ultrasonography (US)-computed tomography (CT)/magnetic resonance (MR) fusion tool guidance. The electrodes will be cooled with saline, and radiofrequency (RF, bipolar mode and switching monopolar mode) will be applied to two electrodes at the same time for about 6 to 30 minutes depending on the tumor size. The temperature will be maintained at 90-100 °C. The RF energy will be delivered by using the 200 watts single generator.

SUMMARY:
To investigate the therapeutic effects and treatment results of radiofrequency ablation using combined bipolar and monopolar energy deliver with twin cooled-wet electrodes for recurrent tumor after locoregional treatment in patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh Class A or B
* chronic hepatitis B or chronic hepatitis C or liver cirrhosis
* presence of recurrent hepatocellular carcinoma (HCC) after locoregional treatment confirmed by pathology or imaging studies including contrast enhanced computed tomography (CT) or magnetic resonance imaging (MRI) according to Liver Imaging Reporting and Data System (LI-RADS) v2018
* single lesion less than or equal to 5 cm, or up to 3 lesions, each greater than less than or equal to 3 cm at the time of locoregional treatment

Exclusion Criteria:

* number of recurrent HCCs, equal or more than 3
* largest recurrent HCC size over 3 cm
* presence of vascular invasion by HCC
* platelet count less than 40,000 per mm3 or International Normalized Ratio (INR) prolongation over 50%
* presence of extrahepatic metastasis

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Local tumor progression rate | 12 months after radiofrequency ablation
  Evaluate local tumor progression by follow-up computed tomography (CT) or magnetic resonance imaging (MRI) with alpha-fetoprotein (AFP) level

SECONDARY OUTCOMES:
Safety margin evaluation | Immediately after radiofrequency ablation
  Evaluate the safety margin around the index tumor on immediate computed tomography (CT)
Technical success rate | 1 month after radiofrequency ablation
  Evaluate technical success defined as complete ablation of the index tumor on 1 month follow-up computed tomography.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea